CLINICAL TRIAL: NCT03696550
Title: A Phase 1, Open-label, Multicenter Study to Determine the Pharmacokinetics and Safety of Intravenous Eravacycline in Children With Suspected or Confirmed Bacterial Infection
Brief Title: A Safety and PK Study of IV Eravacycline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Organization: La Jolla Pharmaceutical Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-434-028
Record Dates: First submitted 2018-09-26; First posted 2018-10-04 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — eravacycline

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Eravacycline (TP-434) intravenous formulation Eravacycline will be administered as a single 60 minute IV infusion according to age.
  Age group (years) Dose (mg/kg) 12 to <18 (Cohort 1) 1.50
  Interventions: Drug: Eravacycline (TP-434)
- Cohort 2 (Experimental): Eravacycline will be administered as a single 60 minute IV infusion according to age.
  Age group (years) Dose (mg/kg) 8 to <12 (Cohort 2) 1.75
  Interventions: Drug: Eravacycline (TP-434)

INTERVENTIONS:
Drug: Eravacycline (TP-434) — Subjects will be stratified by age into 2 cohorts, as follows:
  * Cohort 1: from 12 to <18 years of age (N=8)
  * Cohort 2: from 8 to <12 years of age (N=12 or at least 60% of subjects)
  Other Names: Trade name: Xerava™

SUMMARY:
This is a Phase 1, open-label, multi-center study to determine the pharmacokinetics and safety of intravenous Eravacycline in Children with Suspected or Confirmed Bacterial Infection. Male and Female subjects from 8 to <18 years of age who fulfill the inclusion/exclusion criteria will be enrolled in this study.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single dose study to evaluate PK, safety, and tolerability of IV eravacycline in children with suspected or confirmed bacterial infection who are receiving systemic antibiotic therapy, other than eravacycline. The study design will allow for evaluation of PK and safety of IV eravacycline in a pediatric population at exposures predicted to be comparable to those already studied in adults. The study design is depicted in Figure 1.

Two cohorts defined by age group will be enrolled simultaneously:

* Cohort 1: 12 to <18 years of age (adolescents)
* Cohort 2: 8 to <12 years of age (younger children) Eravacycline will be administered as a single IV dose using the optimum dosage determined from PK-PD modeling and model-based simulations of phase 1, 2, and 3 adult data. Blood samples will be collected for PK analysis at predetermined timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 8 to <18 years of age on the day informed consent (and assent, if applicable) is obtained
2. Written informed consent from parent(s) or other legally authorized representative(s) and informed assent from subject (if age appropriate according to local requirements)
3. Hospitalized, in stable condition, and receiving or plan to receive within 24 hours systemic antibiotic therapy, other than eravacycline, for a suspected or confirmed bacterial infection
4. Likely to survive the current illness
5. In the Investigator's opinion, the subject will require hospitalization for at least 24 hours following administration of the study drug
6. The subject appears to have sufficient intravascular access (peripheral or central) to receive study drug

Exclusion Criteria:

1. Evidence or history of a clinically significant medical condition that may, in the assessment of the Investigator, impair study participation or pose a significant safety risk or diminish the subject's ability to undergo all study procedures and assessments
2. Received an investigational product and/or device within 30 days prior to study drug administration or is currently enrolled in any other clinical study involving an investigational product or any other type of medical treatment judged by the Investigator, in consultation with the Medical Monitor, not to be scientifically or medically compatible with this study
3. History of hypersensitivity to tetracycline antibiotics
4. Prior dosing in this protocol
5. Unlikely to survive at least 48 hours following administration of study drug
6. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol
7. Subject is a child of an employee of the Investigator or study center who has direct involvement in the proposed study or other studies under the direction of the same Investigator or study center, or an immediate family member of the employee or the Investigator, defined as a spouse, parent, child, or sibling, whether biological or legally adopted
8. Breastfeeding females
9. Females of childbearing potential [those with menarche and/or thelarche (beginning of breast development)] and sexually active males who are unwilling or unable to use an acceptable method of contraception
10. Positive pregnancy test in females of childbearing potential
11. Any other circumstance that, in the opinion of the Investigator, would preclude subject participation in the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Assess the Pharmacokinetics (PK) parameters for Cmax, maximum observed plasma concentration | Screening (-2 to 1) to Day 7
  Cmax, maximum observed plasma concentration
Assess the Pharmacokinetics (PK) parameters for AUC0-t, area under the plasma concentration-time curve | Screening (-2 to 1) to Day 7
  AUC0-t, area under the plasma concentration
Assess the Pharmacokinetics (PK) parameters for AUC0-inf, area under the plasma concentration-time curve extrapolated to infinite time | Screening (-2 to 1) to Day 7
  AUC0-inf, area under the plasma concentration-time curve extrapolated to infinite time
Assess the Pharmacokinetics (PK) parameters for AUC0-24, area under the plasma concentration-time curve from time 0 to 24 hours after dose | Screening (-2 to 1) to Day 7
  AUC0-24, area under the plasma concentration-time curve from time 0 to 24 hours after dose
Assess the Pharmacokinetics (PK) parameters for t1/2, elimination half-life | Screening (-2 to 1) to Day 7
  t1/2, elimination half-life
Assess the Pharmacokinetics (PK) parameters for Clast,, last observed plasma concentration | Screening (-2 to 1) to Day 7
  Clast, last observed plasma concentration
Assess the Pharmacokinetics (PK) parameters for CL, systemic clearance | Screening (-2 to 1) to Day 7
  CL, systemic clearance
Assess the Pharmacokinetics (PK) parameters for Vd, volume of distribution | Screening (-2 to 1) to Day 7
  Vd, volume of distribution

SECONDARY OUTCOMES:
Adverse Events | From the time of signing the informed consent form to Day 7
  Assess Adverse Events to assess safety and tolerability
A Directed Physical examination including chest/respiratory | Screening (-2 to 1) to Day 7.
  Changes in Physical examination findings including chest/respiratory
A Directed Physical examination including heart/cardiovascular | Screening (-2 to 1) to Day 7.
  Changes in Physical examination findings including heart/cardiovascular
Vital Signs including blood pressure | Screening (-2 to 1) to Day 7
  Changes in blood pressure
Vital Signs including heart rate | Screening (-2 to 1) to Day 7
  Changes in heart rate
Vital Signs including respiratory rate | Screening (-2 to 1) to Day 7
  Changes in respiratory rate
Vital Signs including body temperature | Screening (-2 to 1) to Day 7
  Changes in body temperature
Safety laboratory results including clinical chemistry | Screening (-2 to 1) to Day 7
  Changes in Clinical laboratory tests including clinical chemistry
Safety laboratory tests including hematology | Screening (-2 to 1) to Day 7
  Changes in Clinical laboratory tests including hematology

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - West Virginia University Hospital, Morgantown, West Virginia